CLINICAL TRIAL: NCT04627870
Title: A Prospective, Multi-center, Randomized Controlled Trial to Evaluate the Safety and Feasibility of Intracranial Drug-coated Balloon Catheter in the Treatment of Intracranial In-stent Restenosis
Brief Title: ACOART Intracranial ISR Pilot:Intracranial DCB in the Treatment of Intracranial In-stent Restenosis
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Acotec Scientific Co., Ltd (Industry)
Collaborators: Beijing Tiantan Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ACOART intracranial ISR pilot
Record Dates: First submitted 2020-11-04; First posted 2020-11-13 (Actual); Last update posted 2024-08-01 (Actual); Status verified 2024-06

CONDITIONS: Intracranial Atherosclerosis; Stroke
Keywords: Intracranial Atherosclerosis; In-stent restenosis; drug coated balloon
MeSH Terms: conditions — Intracranial Arteriosclerosis; Stroke | interventions — Dosage Forms

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- DCB group (Experimental): use drug (paclitaxel) coated balloon to treat intracranial in-stent restenosis
  Interventions: Device: drug (paclitaxel) coated balloon
- PTA group (Active Comparator): use PTA balloon to treat intracranial in-stent restenosis
  Interventions: Device: PTA balloon

INTERVENTIONS:
Device: drug (paclitaxel) coated balloon — use drug (paclitaxel) coated balloon catheter to treat intracranial in-stent restenosis
  Arms: DCB group
Device: PTA balloon — use traditional PTA balloon with NMPA approval of indication for treating intracranial stenosis
  Arms: PTA group

SUMMARY:
The purpose of the study is to evaluate the safety and feasibility of drug coated balloon in treatment of intracranial in-stent restenosis.

DETAILED DESCRIPTION:
This study is a prospective, multi-center, randomized controlled trial using drug coated balloon versus uncoated PTA balloon in treatment of intracranial in-stent restenosis.

ELIGIBILITY:
Inclusion Criteria:

* 18 to 80 years of age
* Confirmed by DSA: in-stent restenosis (ISR) at intracranial segment of internal carotid artery, middle cerebral artery, basilar artery and vertebral artery; ISR is defined as >50% stenosis within or immediately adjacent (within 5 mm) of the implanted stent and >20% absolute luminal loss
* presence of ISR associated ischemic stroke or transient ischemic attacks even with medical treatment and strict control of risk factor
* asymptomatic ISR with severe hypoperfusion in the ISR territories, confirmed by a cerebral blood flow decrease of ≥30% when compared with the perfusion on the contralateral side for anterior circulation lesions or the anterior circulation territory for posterior circulation lesions on CT perfusion, and/or by an American Society of Interventional and Therapeutic Neuroradiology/Society of Interventional Radiology (ASITN/SIR) Collateral Flow Grading System score <3 on DSA.
* the diameter of target vessel is 2.0-4.5mm
* there is only one intracranial ISR lesion per subject
* baseline mRS score ≤2
* Voluntarily participate in this study and sign the informed consent form

Exclusion Criteria:

* Patients with stroke within 2 weeks before procedure;
* any history of brain parenchyma or other intracranial subarachnoid, subdural or extradural hemorrhage in the past 30 days.
* Those who have received thrombolysis within 24 hours before procedure;
* Deterioration of neurological function within 24 hours before procedure (defined as NIHSS score increased by ≥ 4 points over the baseline)
* patients with thrombus in target vessels.
* in addition to ISR lesions, there are other primary intracranial lesions that need endovascular treatment.
* Major surgery (including open femoral, aortic or carotid artery surgery) is planned within the past 30 days or within 90 days.
* patients with renal artery, iliac artery and cardiac coronary artery requiring simultaneous intervention.
* Combined with intracranial tumors, aneurysms or intracranial arteriovenous malformations.
* Cardiac stroke or potential cardiogenic thromboembolism, with any of the following cardiogenic embolism causes: chronic or paroxysmal atrial fibrillation, mitral valve stenosis, mechanical valves, endocarditis, intracardiac thrombus or implant, dilated cardiomyopathy, spontaneous acoustic imaging of the left atrium;
* patients with myocardial infarction within 6 weeks before procedure.
* those who cannot tolerate general anesthesia due to insufficiency of heart, lung and other important organs.
* patients with known severe hepatic and renal dysfunction.
* patients with hemoglobin < 100g / L, platelet count < 100,000 / mm3, INR > 1.5or with uncorrectable factors leading to bleeding.
* patients who cannot receive dual antiplatelet therapy due to existing diseases or who are tested to be tolerant to dual antiplatelet therapy.
* Patients with known severe allergies or contraindications to heparin, paclitaxel, contrast agents and other related intravascular treatment drugs
* current alcohol or drug abuse, uncontrolled severe hypertension (systolic blood pressure > 180mmHg or diastolic blood pressure > 110mmHg).
* Life expectancy < 1 year.
* pregnant or lactating women.
* patients who are unable to complete follow-up due to cognitive, emotional disorders or mental illness.
* Patients who are participating in other drug/device clinical trials and have not completed all follow-ups required by the programme;
* According to the judgement of the investigator, other situations that are not suitable for enrollment

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2021-05-26 (Actual); Primary Completion 2024-12-30 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Target vessel stroke or death event | within 30 days post-procedure
  Target-vessel related stroke (bleeding and ischemia) or death within 30 days postoperatively.

SECONDARY OUTCOMES:
device success rate | assessed during procedure
  The balloon dilatation catheter was able to reach the treated lesion, successfully dilated without rupture, and successfully retreated.
target vessel ischemia stroke event | between 31days and 12months post-procedure
  The incidence of recurrent ischemic stroke in the target vessel supply area 31 days to 12 months after surgery
Cerebral parenchyma hemorrhage, subarachnoid hemorrhage or intraventricular hemorrhage events | between 31 days and 12 months post-procedure
  Any cerebral parenchyma hemorrhage, subarachnoid hemorrhage, or intraventricular hemorrhage confirmed by MRI or CT from 31 days to 12 months post procedure
target vessel death event | between 31 days and 12 months post-procedure
  Target-vessel related death 31 days to 12 months postoperatively
National Institutes of Health Stroke Scale score | at 12 months post-procedure
  National Institutes of Health Stroke Scale score at 12 months postoperatively(0-42, higher scores mean a worse outcome)
Modified Rankin Score score | at 12 months post-procedure
  Modified Rankin Score at 12 months postoperatively(0-5, higher scores mean a worse outcome)

CONTACTS AND LOCATIONS:
Overall Officials: Ning Ma, MD, Principal Investigator — Beijing Tiantan Hospital
Locations (1):
- Beijing Tiantan Hospital, Beijing, China